CLINICAL TRIAL: NCT07048340
Title: The Role of Sleep Restriction Therapy in Cognitive-behavioral Therapy for Insomnia in School-aged Children: A Randomized Controlled Trial
Brief Title: Cognitive-behavioral Therapy for Insomnia in School-aged Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Michal Kahn, Senior lecturer, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0010319-2
Record Dates: First submitted 2025-05-26; First posted 2025-07-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: Insomnia; Pediatric insomnia; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I (Experimental): Families will receive the complete Cognitive Behavioral Therapy for Insomnia protocol (intake session + 4 CBT-I sessions).
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- CBT-I without SRT (Active Comparator): Families will receive the Cognitive Behavioral Therapy for Insomnia protocol (intake session + 4 CBT-I sessions), excluding the Sleep Restriction Therapy (SRT) components.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia without SRT
- Waitlist control (No Intervention): Families will complete the intake session and then be placed on a waitlist and receive CBT-I 5 weeks after baseline.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I intervention will include four 45-60 minute sessions with a clinician. The sessions will include CBT-I components such as sleep psychoeducation, bedtime routines and sleep hygiene, graduated exposure, cognitive restructuring, and SRT in one of the intervention groups. The protocol is based on previous studies of CBT-I for school-aged children.
  Arms: CBT-I
Behavioral: Cognitive Behavioral Therapy for Insomnia without SRT — This intervention will include four 45-60 minute sessions with a clinician. The sessions will include CBT-I components such as sleep psychoeducation, bedtime routines and sleep hygiene, graduated exposure, and cognitive restructuring. Sleep Restriction Therapy will not be included in the intervention. The protocol is based on previous studies that delivered CBT-I to school-aged children.
  Arms: CBT-I without SRT

SUMMARY:
This randomized controlled trial will test the efficacy of CBT-I intervention for school-aged children (7-11 years old) with insomnia. The trial will focus on the role of sleep restriction therapy in treatment. Children will be randomized to one of three groups: (1) CBT-I; (2) CBT-I without SRT; or (3) a waitlist control group. Assessments will occur at baseline, mid-treatment, post-treatment, and a 3-month follow up. Some measures (e.g., child motivation) will also be assessed after each therapy session. Insomnia and sleep-wake patterns will be assessed objectively using actigraphy, and subjectively using sleep diaries, a clinical diagnostic interview, and questionnaires. Parent and child questionnaires will be administered to assess moderators and mediators of treatment outcomes.

DETAILED DESCRIPTION:
Insomnia stands out as the most prevalent sleep disorder in youth, inflicting a range of adverse consequences on both the child and the family. While cognitive-behavioral therapy for insomnia (CBT-I) is considered the first-line treatment, empirical investigations into its efficacy in school-aged children have been scarce. Moreover, the unique contributions and underlying mechanisms of individual treatment components of the CBT-I 'package' remain poorly understood. Sleep Restriction Therapy (SRT) is acknowledged as a core module of CBT-I in adults, presumably driving clinical change via increases in homeostatic sleep pressure that facilitate sleep onset and maintenance. Yet, the incremental benefits of SRT within the context of CBT-I have not been systematically examined. Similarly, the role of two key mechanisms in the CBT-I 'package'-pre-sleep hyperarousal and parental over-accommodation-as mediators of treatment outcome has not been investigated. As for treatment moderators, the frequently encountered lack of motivation among children to engage in therapy poses a notable barrier to effective insomnia treatment, a barrier that SRT may potentially alleviate by offering the appeal of a later bedtime. Given the unique characteristics of insomnia in school-aged children and the prominent role played by parents in etiology and treatment, understanding these processes is pivotal. The proposed dismantling trial is designed to address these issues by rigorously testing the efficacy of CBT-I, including and excluding the SRT module, meticulously examining underlying mechanisms, and determining which variation of the intervention may be more suitable for specific children.

A total of 120 children aged 7-11 with chronic insomnia disorder will be randomized to one of 3 study arms: (1) CBT-I; (2) CBT-I without SRT; or (3) a waitlist control group. Assessments will occur at baseline, mid- treatment, post-treatment, and 3-month follow-up. Insomnia and sleep-wake patterns will be assessed objectively via actigraphy, complemented by parent and child questionnaires, sleep diaries, and a clinical diagnostic interview. Additional factors will be measured, including the child's presleep hyperarousal, separation anxiety, behavioral and emotional problems, as well as parental accommodation, distress and anxiety, and cry tolerance. Some of these factors will be tested as possible mediators (pre-sleep hyperarousal, parental accommodation, child motivation to engage in treatment, and family adherence to treatment) and moderators (parent and child levels of emotional or behavioral problems at baseline) of treatment outcome. Parents' satisfaction with treatment will also be assessed at post-treatment. Participants allocated to the waitlist control group will all receive CBT-I after the 5-week waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 7-11 years
* Parents aged over 18 years
* Child meets the International Classification of Sleep Disorders - Third Edition (ICSD-3) criteria for chronic insomnia disorder with sleep difficulties occurring at least 3 times a week and lasting at least 3 months (Insomnia diagnosis will be determined during a clinical interview).

Exclusion Criteria:

* Child receiving concurrent CBT treatment for sleep or anxiety disorders.
* Child diagnosed with a medical sleep problem (e.g., OSA, RLS)
* Significant health or neurodevelopmental problems (e.g., intellectual disability)
* Current psychotropic medications, or sleep aid medications
* Lack of Hebrew reading and writing
* Total sleep time that is shorter than 6 hours on average per night at baseline

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of child insomnia | Baseline, post-treatment (5 weeks following baseline)
  A structured interview with the child and parents will be conducted at both baseline and post-treatment by a blind clinical assessor. Based on ICSD-3 criteria, children will be diagnosed with chronic insomnia disorder if their sleep difficulties are evident on ≥3 nights per week, persisting for ≥3 months. The interview will additionally address sleep-related behaviors (e.g., reliance on parents for sleep onset), daytime consequences, and differential diagnosis. The clinical diagnosis of insomnia at baseline will serve to confirm that the child qualifies for inclusion in the trial. At post-treatment, the percentage of children no longer meeting the criteria for the disorder will be considered a primary outcome measure.
Child sleep efficiency | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Sleep efficiency will be measured using actigraphy and sleep diaries completed by parents. Sleep efficiency is computed as the percent of total sleep duration out of time in bed (including sleep onset latency and any wakefulness after sleep onset).

SECONDARY OUTCOMES:
Child sleep duration - actigraphic | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Total nighttime sleep duration will be assessed using actigraphy
Child sleep duration - parent reports | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Total nighttime sleep duration will be assessed using sleep diaries completed by parents.
Child number of awakenings - actigraphic | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Number of nighttime awakenings will be assessed using actigraphy.
Child number of awakenings - parent reports | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  The number of nighttime awakenings will be assessed using daily sleep diaries filled by parents.
Number of nights of co-sleeping | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Parents will report in daily sleep diaries whether co-sleeping (sharing a room or bed with the child) occured.
Child sleep related problems | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Sleep behaviors and difficulties will be measured using the Children's Sleep Habit Questionnaire (CSHQ) - a 33-item parent-report measure of sleep behaviors and difficulties.

OTHER OUTCOMES:
Child pre-sleep hyperarousal | Baseline, mid-treatment (3 weeks following baseline), and post-treatment (5 weeks following baseline).
  Presleep Hyperarousal will be assessed using The Pre-Sleep Arousal Survey for Children (PSAS-C), administered to the child by clinicians.
Parental accommodation score (FASS-PR) | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Both parents will complete The Family Accommodation Scale for Sleep- Parent Report (FASS-PR), and a total score will be computed, with higher scores indicating greater parental accommodation.
Parental accommodation - Kalhish Questionnaire | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Both parents will complete The Kalhish Questionnaire, measuring parental cognitions regarding child's anxiety. A total score will be computed, with higher scores indicating more parental cognitions endorsing accommodation.
Child externalizing and internalizing symptoms | Baseline, mid-treatment (3 weeks following baseline), post-treatment (5 weeks following baseline), and follow-up (three months following baseline)
  Child behavioral problems will be assessed using the Strengths and Difficulties Questionnaire (SDQ), parent version.
Parent depression, anxiety, and stress | Baseline and post-treatment (5 weeks following baseline)
  Parent depression, anxiety, and stress symptoms will be assessed using the DASS-21.
Child separation anxiety | Baseline and post treatment (5 weeks following baseline)
  Separation anxiety will be measured using 8 items from the separation anxiety subscale of the Screen for Childhood Anxiety Related Disorders questionnaire (SCARED).
Parental cry tolerance | Baseline
  Parents will undergo the Intervention Delay to Infant Crying Video (IDICV), which measures response time to a crying baby.
  The IDICV includes a presentation of a 2-min video clip of a 6-month-old baby playing on a carpet who then starts crying (after 10s), with a gradual increase in crying intensity and visual distress signs. Directions prior to the video presentation include that the parents of the baby are trying to ignore some of his crying to allow him to calm down by himself, and participants are asked to decide when they feel that it is absolutely necessary to intervene.
Treatment adherence - parent reports | After each of the 4 therapy sessions, including session 1 (1 week after baseline), session 2 (2 weeks after basline), 3 (3 weeks after baseline), and 4 (5 weeks after baseline).
  Parents will complete a questionnaire regarding their adherence to the treatment protocol after every session. Parent ratings will be averaged to create a parental adherence score, with higher scores indicating higher adherence to treatment.
Treatment adherence - therapist reports | After each of the 4 therapy sessions, including session 1 (1 week after baseline), session 2 (2 weeks after basline), 3 (3 weeks after baseline), and 4 (5 weeks after baseline).
  Therapists will evaluate the family's adherence to the treatment protocol after every session. Ratings will be averaged to create a family adherence score, with higher scores indicating higher adherence to treatment.
Child motivation for treatment - child reports | After each of the 4 therapy sessions, including session 1 (1 week after baseline), session 2 (2 weeks after basline), 3 (3 weeks after baseline), and 4 (5 weeks after baseline).
  Children will answer modified questions from the Child Motivation Scale, administered by the clinician. Ratings will be averaged to create a child motivation score, with higher scores indicating higher motivation for treatment.
Child motivation for treatment - therapist reports | After each of the 4 therapy sessions, including session 1 (1 week after baseline), session 2 (2 weeks after basline), 3 (3 weeks after baseline), and 4 (5 weeks after baseline).
  Therapists will also assess the motivation of the family (child and parents) on questionnaire items. Ratings will be averaged to create a family motivation score, with higher scores indicating higher motivation for treatment.
Treatment satisfaction - parent reports | After each of the 4 therapy sessions, including session 1 (1 week after baseline), session 2 (2 weeks after basline), 3 (3 weeks after baseline), and 4 (5 weeks after baseline).
  Parents will answer questions regarding their satisfaction with the treatment and their relationship with the clinician. Ratings will be averaged to create a total satisfaction score, with higher scores indicating higher satisfaction from treatment.
Treatment satisfaction - child reports | After each of the 4 therapy sessions, including session 1 (1 week after baseline), session 2 (2 weeks after basline), 3 (3 weeks after baseline), and 4 (5 weeks after baseline).
  Children will answer questions regarding their satisfaction with the treatment after each session. Their ratings will be averaged to create a total satisfaction score, with higher scores indicating higher satisfaction from treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data upon reasonable request, including baseline demographic and clinical characteristics (e.g., age, gender, diagnosis, symptom severity at baseline), intervention assignment, and primary and secondary outcome measures. Data will be fully anonymized to protect participant confidentiality before sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From June 2025 Until 7 years after study completion (anticipated December 2029)
Access Criteria: Qualified researchers affiliated with academic or clinical institutions will be able to request access to the de-identified individual participant data (IPD) and supporting documentation. Requests for access will be reviewed on a case-by-case basis to ensure appropriate use and compliance with ethical and legal standards. Interested researchers can submit a data request to the corresponding author via email, including a brief proposal outlining the intended use and planned analyses. A data sharing agreement will be required prior to access. Data will be shared electronically via secure institutional file transfer systems.
URL: https://osf.io